CLINICAL TRIAL: NCT02126033
Title: Telomeres Parameters in Celiac Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, ido laish, physician in gastroenterlogy institute, Meir Medical Center
Model: Parallel | Purpose: Basic Science
Other Study IDs: 1234
Record Dates: First submitted 2014-04-27; First posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Celiac Disease
Keywords: celiac; telomere; telomerase
MeSH Terms: conditions — Celiac Disease

ARMS (1):
- celiac disease (Experimental)
  Interventions: Procedure: take blood samples

INTERVENTIONS:
Procedure: take blood samples

SUMMARY:
Celiac disease is an autoimmune process that causes destructive changes in the epithel of the small bowel and it is also a pre-malignant state (e.g lymphoma). The aim of the study is to examine telomere length and other parameters of genetic instability from peripheral blood lymphocytes of patients with celiac disease compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* patients with celiac disease

Exclusion Criteria:

* known malignancy
* cannot sign informed consent
* under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
telomere length | at entry, after 6 months of gluten-free diet